CLINICAL TRIAL: NCT02546414
Title: Platelet Count（PC）/Spleen Diameter(SD) Ratio to Predict the Variceal Haemorrhage in HBV Cirrhotic Patients in China
Status: Completed | Type: Observational
Sponsor: RenJi Hospital (Other)
Responsible Party: Principal Investigator, Shengliang Chen, MD, RenJi Hospital
Other Study IDs: RJLIJINHUI-2015
Record Dates: First submitted 2015-08-26; First posted 2015-09-10 (Estimated); Last update posted 2015-09-10 (Estimated); Status verified 2015-09

CONDITIONS: Platelet Count/Spleen Diameter Ratio; Child-Pugh Classification
Keywords: Platelet count/spleen diameter ratio; China
MeSH Terms: interventions — Platelet Count

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Esophageal varices haemorrhage group: HBV hepatic cirrhosis with first esophageal varices haemorrhage were included and stratified using their Child-Pugh score. The platelet count were evaluated, and ultrasound was used to measure the longest diameter of the spleen. The platelet count(PC)/spleen diameter (SD)ratio was calculated and analyzed to determine whether it can predict the variceal haemorrhage. Upper gastrointestinal endoscopy was used as the gold standard.
  Interventions: Other: Platelet count/spleen diameter ratio
- no haemorrhage but esophageal varice presence: HBV hepatic cirrhosis with no esophageal varices haemorrhage were included and upper gastrointestinal endoscopy were validate.They also stratified using their Child-Pugh score. The platelet count and longest diameter of the spleen were evaluated, The PC/SD ratio was calculated and analyzed to determine whether it can predict the variceal presence.
  Interventions: Other: Platelet count/spleen diameter ratio
- no esophageal varice but cirrhotic: HBV hepatic cirrhosis with no esophageal varices were included and also validated by upper gastrointestinal endoscopy.They stratified using their Child-Pugh score. The platelet count and longest diameter of the spleen were evaluated,The PC/SD was calculated and analyzed to determine whether it can predict the variceal absence .
  Interventions: Other: Platelet count/spleen diameter ratio

INTERVENTIONS:
Other: Platelet count/spleen diameter ratio — Platelet count were evaluated by complete blood count, and ultrasound was used to measure the longest diameter of the spleen.The platelet count/spleen diameter ratio was calculated
  Other Names: PC/SD ratio

SUMMARY:
To validate the PC/SD ratio to be used to predict the variceal haemorrhage in Chinese patients with hepatitis B virus (HBV)-associated hepatic cirrhosis.

DETAILED DESCRIPTION:
Esophageal variceal bleeding remains the leading cause of acute mortality in patients with cirrhosis. Using noninvasive parameters for high-risk variceal haemorrhage may reduce the need for endoscopies. The ratio of platelet count/diameter of the spleen (PC/SD ratio) is the principal noninvasive predictor of esophageal varices. This was an analytical cross-sectional study to validate the diagnostic test for HBV hepatic cirrhosis and was performed between January 2013 and August 2015. This study is to validate the PC/SD ratio to identification of those patients with high bleeding risk and selection for prophylactic treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of HBV hepatic cirrhosis

Exclusion Criteria:

* Patients with hepatocellular carcinoma,
* use of medications for the primary prophylaxis of variceal bleeding,
* history of esophageal variceal bleeding,
* alcohol consumption within the admission and a history of ligation,
* sclerotherapy, and/or
* portal hypertension surgery

Ages: 45 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HBV cirrhotic patients in China
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2013-01; Primary Completion 2015-07 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Platelet count/spleen diameter ratio | up to 2.5 years
  This was an analytical cross-sectional study to validate the diagnostic test for HBV hepatic cirrhosis and was performed between January 2013 and August 2015

SECONDARY OUTCOMES:
Child-Pugh score. | up to 2.5 years
  This was an analytical cross-sectional study to validate the diagnostic test for HBV hepatic cirrhosis and was performed between January 2013 and August 2015

CONTACTS AND LOCATIONS:
Locations (1):
- Renji Hospital, Shanghai, Shanghai Municipality, China